CLINICAL TRIAL: NCT03759145
Title: The Jintronix Interactive System for Upper Extremity Rehabilitation Training Post Stroke: A Pilot Study
Brief Title: The Jintronix Interactive System for Upper Extremity Rehabilitation Training Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Dahlia Kairy, Associate professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRIR-795-0113
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Stroke
Keywords: virtual reality; exergame; stroke rehabilitation
MeSH Terms: conditions — Stroke | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm, usual rehabilitation + Jintronix exergame (Experimental): On top of the usual out-patient rehabilitation sessions planned for the participant, participants attend sessions to use the Jintronix system for up 30 minutes up to 3 times per week
  Interventions: Other: Exergame
- Control group (Other): Participants continue their prescribed rehabilitation sessions
  Interventions: Other: usual care

INTERVENTIONS:
Other: Exergame — Participants use exergame with the therapist in the rehabilitation center. Several games are available, the therapist adjusts the choice of game and level of difficulty according to the participant's abilities and interests.
  Arms: Intervention arm, usual rehabilitation + Jintronix exergame
Other: usual care — participants continued their planned rehabilitation sessions
  Arms: Control group

SUMMARY:
Stroke is a leading cause of death and disability worldwide.Hemiplegia, weakness of one side of the body, is a common consequence of stroke that can lead to significant functional impairments. Loss of arm function occurs in up to 85% of stroke survivors. The impact of arm-related limitations on activities of daily living, leisure activities or work is significant as the arm plays a central role in a person's life from the ability to perform basic activities of daily life to carrying out family and social roles. Guidelines indicate that rehabilitation can improve upper extremity (UE) motor control and functional status post stroke. Virtual reality (VR) and computer games are recent technologies that, as they become more accessible and affordable,are increasingly being used in rehabilitation to allow patients to engage in repetitive practice of specific tasks. A number of published reviews and meta-analyses have examined the use of VR and video games for post-stroke rehabilitation, focusing on or including UE rehabilitation. The authors agree that there is limited but promising findings that VR and video-games, when combined with traditional rehabilitation, have a positive impact on recovery post-stroke.

DETAILED DESCRIPTION:
The goal of the study is to assess the feasibility, safety, and acceptability of the Jintronix system, as well as provide preliminary evidence regarding the clinical efficacy for post-stroke rehabilitation.This is a pilot parallel randomised single-blinded controlled trial, with patients who have had a stroke randomly allocated to one of two groups: (1) usual rehabilitation services and additional training with Jintronix system (treatment group) or (2) usual rehabilitation services only (control group).

ELIGIBILITY:
Inclusion Criteria:

* having had an ischemic or hemorrhagic stroke for the first time;
* having residual mild to moderate UE impairment (score 3-6 on the Chedoke-McMaster arm component, as long as exergames can be played);
* being in subacute stage (within 6 months post-stroke);
* receiving usual out-patient rehabilitation services at one of the two selected rehabilitation sites, located in the greater Montreal area in Canada.

Exclusion Criteria:

* being medically unstable;
* having severe cognitive or communication deficits;
* having visual impairments limiting use of the exergame;
* having any medical contraindication for shoulder movements;
* having severe balance deficits limiting sitting safely independently;
* having previous upper limb impairment limiting potential recovery;
* having any other impairment that limited use of the exergame.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
number of sessions (feasibility) | 4 week period
  number of sessions the participant used the system during the study period
duration of sessions | 4 week period (ongoing)
  the average duration of sessions (minutes)
time spent by therapist assisting the participant | 4 week period (ongoing)
  time during the sessions that the therapist spent assisting the participant (minutes)
time spent on each exergame | 4 week period (ongoing)
  the time spent on each exergame (minutes)
adverse event (counts) | 4 week period (ongoing)
  occurrence of adverse events such as falls, motion sickness, dizziness and headaches
adverse event (borg exertion scale, self-reported scale 6-20, (Borg Exertion Scale scored from 6-20, no exertion to maximal exertion) | 4 week period (ongoing)
  exertion after playing the exergame reported using the Borg Exertion Scale
adverse event (pain self reported on visual analog scale 0-10) | 4 week period (ongoing)
  pain after playing the exergame reported using visual analog scale 0-10, 0 is no pain, 10 is the worse pain imaginable.
Stroke-specific measure of quality of life - Stroke Impact Scale | 4 week period (per-post)
  Stroke Impact Scale is a questionnaire of the impact that the stroke is having on function, mood, emotional status, total score 0-100, with with higher scores indicating better self-reported health.
upper limb function assessed using the Motor Activity Log | 4 week period (per-post)
  The Motor Activity Log is a questionnaire that the participant completes reporting how much the impaired upper limb is used for various daily tasks, each task is scored from 0-5 (ordinal scale, 0=do not use arm - 6=use as much as before), total score is mean of the scores.
upper limb function assessed using the Box and Block test | 4 week period (per-post)
  upper limb function is assessed using the box and block test where participants are timed while picking up and placing wooden cubes
upper limb motor control assessed using the Fugl-Meyer Assessment-upper extremity | 4 week period (per-post)
  Upper limb motor control is assessed using a valid and reliable outcome, measure consisting of tasks to be performed by the participant, scores between 0-66, higher scores indicating better motor control.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No